CLINICAL TRIAL: NCT07179965
Title: Nutrition, Meal Regularity and Quality of Life in Inflammatory Bowel Disease
Acronym: Public health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Elif Nur Özen, Research Assistant, Istinye University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IstinyeElif1; No funding (Other: No funding)
Record Dates: First submitted 2025-09-04; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Inflammatory Bowel Disease (IBD); Inflammation; Nutrition; Diet Habits; Gastrointestinal
Keywords: Inflammatory Bowel Disease; Nutrition; Diet; Meal regularity
MeSH Terms: conditions — Inflammatory Bowel Diseases; Inflammation; Feeding Behavior | interventions — Observation

STUDY DESIGN:
Intervention Model Description: Cross sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inflammatory Bowel Disease patients (Other)
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — IBD patients

SUMMARY:
Aims: This study aimed to assess nutritional status, dietary habits, meal patterns, gastrointestinal symptoms, quality of life, and depression in Inflammatory Bowel Disease (IBD) patients.

Methods: Data were collected at a university hospital using the 24-Hour Dietary Recall, IBD Quality of Life Questionnaire, Beck Depression Inventory II, and the Gastrointestinal Symptom Rating Scale.

DETAILED DESCRIPTION:
Inflammatory Bowel Disease (IBD), which is divided into Ulcerative Colitis and Crohn's Disease, is influenced by various environmental factors, including nutrition, and significantly reduces the quality of life. This study included 50 individuals aged 18-75 who were diagnosed with Inflammatory Bowel Disease by a physician, had no communication difficulties, and were able to make their own food choices. The study aimed to evaluate the nutritional status, dietary habits, food consumption frequencies, and meal patterns of the patients and, based on these data, to determine their gastrointestinal symptoms, quality of life, and depression status. The study commenced with ethical approval and was conducted with patients at the Gastroenterology Clinic of Istanbul University Cerrahpaşa Medical Faculty Hospital between August 2023 and September 2023. The research is cross-sectional. Data were collected using the General Information and Nutrition Behaviors Questionnaire, Food Frequency Questionnaire, 24-Hour Dietary Recall, Inflammatory Bowel Disease Quality of Life Questionnaire, Beck Depression Inventory, and Gastrointestinal Symptom Rating Scale.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria required the ability to communicate effectively and make independent dietary choices.

Exclusion Criteria:

* Individuals with psychiatric disorders, or those who were pregnant or breastfeeding, were excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
Weight | Baseline
  kg
Height | Baseline
  cm
24-Hour Dietary Recall | 24-Hour Dietary Recall
IBD Quality of Life Questionnaire | Baseline
  To assess quality of life, the "Inflammatory Bowel Disease Quality of Life Questionnaire," consisting of 36 items and evaluating systemic symptoms, bowel symptoms, functional impairment, social impairment, and emotional functioning, was used. A higher score is associated with better quality of life.
Beck Depression Inventory II | Baseline
  The Beck Depression Inventory-II (BDI-II), a 21-item self-report questionnaire assessing characteristic attitudes and symptoms of depression, was administered at baseline (single time point, at questionnaire administration). Each item is scored on a 4-point scale (0-3), with a total score range of 0-63. Higher scores indicate greater severity of depression, classified as minimal (0-13), mild (14-19), moderate (20-28), and severe (29-63).
Gastrointestinal Symptom Rating Scale | Baseline
  The Gastrointestinal Symptom Rating Scale (GSRS), a 15-item questionnaire comprising five subcategories (abdominal pain, indigestion, diarrhea, constipation, and reflux), was administered at baseline (single time point, at questionnaire administration). Each item is scored on a 7-point Likert scale (1-7), yielding a total score range of 15-105, with higher scores indicating more severe gastrointestinal symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alavinejad P, Hashemi SJ, Behl N, Hormati A, Elbasuny A, Daryani NE, Modarres MP, Arshadzadeh M, Panahande S, Hang DV, Mahros AM, Parsi A, Javaherizadeh H, Rehman A, Pawlak KM, Ahmadi M, Ahmed MH, Farsi F, Arefi M, Quadri A, Tran QT, Alborzi F, Amin Alavi SM, Cheraghian B, Ramezani E, Gouda MF, Saadati B, Quadri AA, Hirani R, Maher M, Ghoneem E. Inflammatory bowel disease evolution in the past two decades: a chronological multinational study. EClinicalMedicine. 2024 Mar 15;70:102542. doi: 10.1016/j.eclinm.2024.102542. eCollection 2024 Apr. PMID 38525407